CLINICAL TRIAL: NCT00922272
Title: A Phase 2, Multicenter Study With Open-label & Randomized Double-blind Placebo-controlled Withdrawal Phases to Evaluate the Efficacy, Safety, & Tolerability of SPD489 in Adults With Schizophrenia & Predominant Negative Symptoms Who Are Clinically Stable & Taking Stable Doses of Atypical Antipsychotic Medication
Brief Title: Efficacy, Safety, and Tolerability of SPD489 in Adults With Schizophrenia and Predominant Negative Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-204
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Results first posted 2012-02-20 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Schizophrenia and Predominant Negative Symptoms
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPD489 (Lisdexamfetamine dimesylate) (Experimental)
  Interventions: Drug: SPD489 (lisdexamfetamine dimesylate)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo matching SPD489 (lisdexamfetamine dimesylate)

INTERVENTIONS:
Drug: SPD489 (lisdexamfetamine dimesylate) — oral, 20, 30, 40, 50, 60, or 70 mg once daily
  Other Names: Vyvanse
  Arms: SPD489 (Lisdexamfetamine dimesylate)
Drug: Placebo matching SPD489 (lisdexamfetamine dimesylate) — oral, once daily
  Arms: Placebo

SUMMARY:
To explore the efficacy of SPD489, as adjunctive therapy to a stable dose of atypical antipsychotic medication, on negative symptoms in adult subjects with clinically stable schizophrenia and predominant negative symptoms, as measured by the Scale for the Assessment of Negative Symptoms (SANS).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55
* Clinically stable Schizophrenia and predominant negative symptoms
* Taking a stable dose of antipsychotic medication

Exclusion Criteria:

* Clinically notable positive symptoms defined by PANSS

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2009-09-14 (Actual); Primary Completion 2011-01-20 (Actual); Study Completion 2011-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (27):
- United States (27):
  - K&S Professional Research Services, Little Rock, Arkansas
  - South Coast Clinical Trials, Anaheim, California
  - Omega Clinical Trials, Anaheim, California
  - Clinical Innovations, Costa Mesa, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Apostle Clinical Trials, Inc., Long Beach, California
  - Excell Research, Inc., Oceanside, California
  - Southcoast Clinical Trials, San Bernardino, California
  - CNRI San Diego & Los Angeles, San Diego, California
  - Affiliated Research Institute, San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Accurate Clinical Trials, Kissimmee, Florida
  - Behavioral Clinical Research, INC, Lauderhill, Florida
  - Segal Institute for Clinical Research (Miami), North Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Comprehensive NeuroScience, Atlanta, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - J. Gary Booker, MD, APMC, Shreveport, Louisiana
  - CRI Worldwide, LLC., Willingboro, New Jersey
  - Advanced Bio-Behavioral Sciences, Elmsford, New York
  - Comprehensive Neuroscience, Inc., Hollis, New York
  - University of Cincinnati, Cincinnati, Ohio
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Community Clinical Research, Inc., Austin, Texas
  - University Hills Clinical Research, Irving, Texas

REFERENCES:
- [Result] Lasser RA, Dirks B, Nasrallah H, Kirsch C, Gao J, Pucci ML, Knesevich MA, Lindenmayer JP. Adjunctive lisdexamfetamine dimesylate therapy in adult outpatients with predominant negative symptoms of schizophrenia: open-label and randomized-withdrawal phases. Neuropsychopharmacology. 2013 Oct;38(11):2140-9. doi: 10.1038/npp.2013.111. Epub 2013 May 8. PMID 23756608
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a 10-week Open-label Phase (7-week Dose Optimization Period and a 3-week Dose maintenance Period) in which subjects received 20 to 70 mg of SPD489 (Lisdexamfetamine dimesylate) once-daily. They were then randomized into the Double-Blind Phase receiving either their optimal dose of SPD489 or placebo once-daily for 4 weeks.
Groups:
- SPD489: The study consisted of a 10-week Open-label Phase (7-week Dose Optimization Period and a 3-week Dose maintenance Period) in which subjects received 20, 30, 40, 50, 60 or 70 mg of adjunctive SPD489 (Lisdexamfetamine dimesylate) once-daily to a stable dose of atypical antipsychotic medication. They were then randomized into the Double-Blind Phase receiving either their optimal dose of adjunctive SPD489 or placebo once-daily for 4 weeks to a stable dose of atypical antipsychotic medication.
- Placebo: Subjects received placebo once-daily for 4 weeks during the Double-blind Phase to a stable dose of atypical antipsychotic medication.
Period: Open-label Phase
Arm/Group | SPD489 | Placebo
Started | 92 | 0
Completed | 69 | 0
Not Completed | 23 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 11 | 0
Not completed — Failure to meet randomization criteria | 1 | 0
Not completed — Withdrawal criteria met | 5 | 0
Period: Double-blind Phase
Arm/Group | SPD489 | Placebo
Started | 34 | 35
Completed | 27 | 29
Not Completed | 7 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal criteria met | 1 | 1
Not completed — Noncompliance | 1 | 1
Not completed — Positive urine drug screen | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall: Constitutes all subjects contained in the Safety Analysis Set defined as all subjects who took at least 1 dose of open-label investigational product and for whom at least 1 follow-up safety assessment was made.
Arm/Group | Overall
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (9.11)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0
  Between 18 and 55 years | 92
  >55 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 62
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 92

OUTCOME MEASURES:

1. Primary Outcome: Change From Open-label Baseline in Modified Scale for the Assessment of Negative Symptoms (SANS-18) Total Score at Week 10 Open-label Phase, Last Observation Carried Forward (LOCF)
Description: The SANS was modified by eliminating the global and attention items; the score of the remaining non-global items is referred to as the SANS-18 total score. Each of the 18-items is scored on a scale from 0 (not at all) to 5 (severe) with a total scoring range of 0 to 90. Higher scores indicate more impairment.
Time Frame: Open-label Baseline and Week 10 Open-label Phase
Population: Open-label Phase Full Analysis Set (FAS) defined as all enrolled subjects who took at least 1 dose of the investigational product and had 1 primary efficacy assessment after baseline in the Open-label Phase.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- SPD489 (Open-label Phase): A 10-week Open-label Phase (7-week Dose Optimization Period and a 3-week Dose maintenance Period) in which subjects received 20, 30, 40, 50, 60 or 70 mg of adjunctive SPD489 (Lisdexamfetamine dimesylate) once-daily to a stable dose of atypical antipsychotic medication.
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 92
Units on a scale | -12.9 (10.04)
Statistical Analysis 1: Comparison: SPD489 (Open-label Phase); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Percent of Participants In Open-label Phase Who Were SANS-18 Responders at Week 10 Open-label Phase
Description: Response is defined as reduction in total SANS score of greater than or equal to 20%. The SANS was modified by eliminating the global and attention items; the score of the remaining non-global items is referred to as the SANS-18 total score. Each of the 18-items is scored on a scale from 0 (not at all) to 5 (severe) with a total scoring range of 0 to 90. Higher scores indicate more impairment.
Time Frame: Week 10 Open-label Phase
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 70
Percent of participants | 52.9

3. Primary Outcome: Change From Double-blind Randomization Baseline in SANS-18 Total Score at Week 4 Double-blind Phase, Termination Observation Carried Forward (TOCF)
Description: as for outcome 1
Time Frame: Double-blind Randomization Baseline and Week 4 Double-blind Phase
Population: Randomized Evaluable Set (RES) defined as all randomized subjects who were responders (Response is defined as reduction in total SANS score of greater than or equal to 20%) at the Double-blind Randomization and had SANS-18 total scores at week 4 of the Double-blind Phase or the early termination visit.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- SPD489 (Double-blind Phase): Subjects receive optimal dose (20, 30, 40, 50, 60 or 70 mg) of adjunctive SPD489 (Lisdexamfetamine dimesylate) once-daily for 4 weeks to a stable dose of atypical antipsychotic medication.
- Placebo (Double-blind Phase): Subjects receive placebo once-daily for 4 weeks to a stable dose of atypical antipsychotic medication.
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 15 | 20
Units on a scale | 4.5 (2.14) | 2.2 (1.85)
Statistical Analysis 1: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Test type: Superiority or Other; p = 0.4182, ANCOVA; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-3.4 to 8.1]

4. Secondary Outcome: Percent of Participants In Double-blind Phase Who Maintained SANS-18 Response at Week 4 Double-blind Phase
Description: as for outcome 2
Time Frame: Week 4 Double-blind Phase
Population: RES
Measure: Number; unit: Percent of participants
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 14 | 17
Percent of participants | 71.4 | 82.4
Statistical Analysis 1: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Test type: Superiority or Other; p = 0.6705, Fisher Exact

5. Secondary Outcome: Change From Open-label Baseline in SANS Global Scores at Week 10 Open-label Phase
Description: The SANS assesses 5 symptom complexes to rate the negative symptoms of subjects. Each of the 18-items is scored on a scale from 0 (not at all) to 5 (severe) with a total scoring range of 0 to 90. Higher scores indicate more impairment.
Time Frame: Open-label Baseline and Week 10 Open-label Phase
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 70
Units on a scale
  Affective Flattening | -0.9 (0.80)
  Alogia | -0.9 (0.65)
  Avolition-Apathy | -0.5 (0.81)
  Anhedonia-Asociality | -0.7 (0.77)
  Attention | -0.7 (0.80)
Statistical Analysis 1: Comparison: SPD489 (Open-label Phase); Affective Flattening; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: SPD489 (Open-label Phase); Alogia; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: SPD489 (Open-label Phase); Avolition-Apathy; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: SPD489 (Open-label Phase); Anhedonia-Asociality; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: SPD489 (Open-label Phase); Attention; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Change From Double-blind Randomization Baseline in SANS Global Scores at Week 4 Double-blind Phase
Description: as for outcome 5
Time Frame: Double-blind Randomization Baseline and Week 4 Double-blind Phase
Population: RES
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 14 | 17
Units on a scale
  Affective Flattening | 0.2 (0.17) | 0.2 (0.15)
  Alogia | 0.5 (0.21) | 0.0 (0.19)
  Avolition-Apathy | 0.2 (0.16) | 0.1 (0.15)
  Anhedonia-Asociality | 0.3 (0.18) | 0.1 (0.16)
  Attention | 0.4 (0.18) | 0.3 (0.17)
Statistical Analysis 1: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Affective Flattening; Test type: Superiority or Other; p = 0.8771, ANCOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.5]
Statistical Analysis 2: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Alogia; Test type: Superiority or Other; p = 0.0584, ANCOVA; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [0.0 to 1.1]
Statistical Analysis 3: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Avolition-Apathy; Test type: Superiority or Other; p = 0.5215, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.6]
Statistical Analysis 4: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Anhedonia-Asociality; Test type: Superiority or Other; p = 0.4835, ANCOVA; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.3 to 0.7]
Statistical Analysis 5: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Attention; Test type: Superiority or Other; p = 0.5723, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.4 to 0.7]

7. Secondary Outcome: Change From Open-label Baseline in Positive and Negative Syndrome Scale (PANSS) Scores at Week 10 Open-label Phase, LOCF
Description: The PANSS is a validated measure that evaluates the presence, absence, and severity of 30 symptoms of schizophrenia including both positive and negative symptoms and general psychopathology. Each of the 30-items are rated on a scale of 1 (absent) to 7 (extreme) with a total scoring range of 30 to 210. Higher scores indicate more impairment.
Time Frame: Open-label Baseline and Week 10 Open-label Phase
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 92
Units on a scale
  Positive subscale | -1.0 (2.23)
  Negative subscale | -4.8 (4.01)
  General Psychopathology subscale | -4.0 (5.11)
Statistical Analysis 1: Comparison: SPD489 (Open-label Phase); Positive subscale; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: SPD489 (Open-label Phase); Negative subscale; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: SPD489 (Open-label Phase); General Psychopathology subscale; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

8. Secondary Outcome: Change From Double-blind Randomization Baseline in PANSS Scores at Week 4 Double-blind Phase, TOCF
Description: as for outcome 7
Time Frame: Double-blind Randomization Baseline and Week 4 Double-blind Phase
Population: Randomized FAS defined as all subjects who received randomized investigational product and had a SANS-18 total scores at week 4 or at the early termination visit.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 34 | 35
Units on a scale
  Positive subscale | 0.5 (0.31) | -0.1 (0.31)
  Negative subscale | 0.9 (0.46) | -0.1 (0.45)
  General Psychopathology subscale | 0.9 (0.78) | -0.9 (0.77)
Statistical Analysis 1: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Positive subscale; Test type: Superiority or Other; p = 0.1975, ANCOVA; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.3 to 1.5]
Statistical Analysis 2: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Negative subscale; Test type: Superiority or Other; p = 0.1228, ANCOVA; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-0.3 to 2.3]
Statistical Analysis 3: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); General Psychopathology subscale; Test type: Superiority or Other; p = 0.1115, ANCOVA; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-0.4 to 3.9]

9. Secondary Outcome: Percent of Participants With Clinical Global Impression - Severity of Illness (CGI-S) at Open-label Baseline
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill)
Time Frame: Open-label Baseline
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 92
Percent of participants
  Normal, not at all ill | 0
  Borderline mentally ill | 0
  Mildly ill | 29.3
  Moderately ill | 55.4
  Markedly ill | 14.1
  Severely ill | 1.1
  Among the most extremely ill | 0

10. Secondary Outcome: Percent of Participants With CGI-S at Week 10 Open-label Phase
Description: as for outcome 9
Time Frame: Week 10 Open-label Phase
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 70
Percent of participants
  Normal, not at all ill | 0
  Borderline mentally ill | 2.9
  Mildly ill | 54.3
  Moderately ill | 38.6
  Markedly ill | 4.3
  Severely ill | 0
  Among the most extremely ill | 0

11. Secondary Outcome: Percent of Participants With CGI-S at Double-blind Randomization Baseline
Description: as for outcome 9
Time Frame: Double-blind Randomization Baseline
Population: Randomized FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 34 | 35
Percent of participants
  Normal, not at all ill | 0 | 0
  Borderline mentally ill | 2.9 | 2.9
  Mildly ill | 50.0 | 60.0
  Moderately ill | 38.2 | 37.1
  Markedly ill | 8.8 | 0
  Severely ill | 0 | 0
  Among the most extremely ill | 0 | 0

12. Secondary Outcome: Percent of Participants With CGI-S at Week 4 Double-blind Phase
Description: as for outcome 9
Time Frame: Week 4 Double-blind Phase
Population: Randomized FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 29 | 29
Percent of participants
  Normal, not at all ill | 0 | 0
  Borderline mentally ill | 3.4 | 13.8
  Mildly ill | 34.5 | 69.0
  Moderately ill | 48.3 | 13.8
  Markedly ill | 13.8 | 3.4
  Severely ill | 0 | 0
  Among the most extremely ill | 0 | 0

13. Secondary Outcome: Percent of Participants With Improvement on Clinical Global Impression - Change (CGI-C) at Week 10 Open-label Phase
Description: CGI-C permits a global evaluation of the change of the subject's overall schizophrenia condition over time. It consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: Open-label Phase Week 10
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 70
Percent of participants | 30.0

14. Secondary Outcome: Percent of Participants With Improvement on CGI-C at Week 4 Double-blind Phase
Description: as for outcome 13
Time Frame: Double-blind Phase Week 4
Population: Randomized FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 29 | 29
Percent of participants | 17.2 | 27.6

15. Secondary Outcome: Change From Open-label Baseline in the Brief Assessment of Cognition in Schizophrenia (BACS) Total Score at Week 10 Open-label Phase
Description: BACS measures attention and speed of processing, and the test score is the total number correct. The measure of the test is the number of correct numerals where subjects write numerals 1-9 as matches to nonmeaningful symbols on a response sheet for 90 seconds, based upon a key provided to them.
Time Frame: Open-label Baseline and week 10 Open-label Phase
Population: FAS
Measure: Mean (Standard Deviation); unit: correct numerals
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 73
correct numerals | 2.3 (8.92)
Statistical Analysis 1: Comparison: SPD489 (Open-label Phase); Test type: Superiority or Other; p = 0.0307, t-test, 2 sided

16. Secondary Outcome: Change From Double-blind Randomization Baseline in BACS Total Score at Week 4 Double-blind Phase
Description: as for outcome 15
Time Frame: Double-blind Randomization Baseline and Week 4
Population: Randomized FAS
Measure: Least Squares Mean (Standard Error); unit: correct numerals
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 32 | 31
correct numerals | 0.1 (1.19) | -2.7 (1.21)
Statistical Analysis 1: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Test type: Superiority or Other; p = 0.1072, ANCOVA; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-0.6 to 6.2]

17. Secondary Outcome: Change From Open-label Baseline in Letter-Number Span Test (LNS) Total Score at Week 10 Open-label Phase
Description: LNS is a test of verbal working memory. Subjects are presented with a sequence of numbers and letters aurally and then asked to tell the rater the numbers first from lowest to highest followed by the letters in alphabetical sequence. The measure is the number of correct sequences.
Time Frame: Open-label Baseline and week 10 Open-label Phase
Population: FAS
Measure: Mean (Standard Deviation); unit: correct sequences
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 73
correct sequences | 0.8 (7.72)
Statistical Analysis 1: Comparison: SPD489 (Open-label Phase); Test type: Superiority or Other; p = 0.3660, t-test, 2 sided

18. Secondary Outcome: Change From Double-blind Randomization Baseline in LNS Total Score at Week 4 Double-blind Phase
Description: as for outcome 17
Time Frame: Double-blind Randomization Baseline and Week 4
Population: Randomized FAS
Measure: Least Squares Mean (Standard Error); unit: correct sequences
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 32 | 31
correct sequences | -0.1 (1.26) | 1.3 (1.28)
Statistical Analysis 1: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Test type: Superiority or Other; p = 0.4347, ANCOVA; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-5.0 to 2.2]

19. Secondary Outcome: Change From Open-label Baseline in Hopkins Verbal Learning Test - Revised (HVLT-R) Total Score at Week 10 Open-label Phase
Description: HVLT-R measures verbal learning. Test scores are the total number of words recalled correctly over 3 trials. The test consists of 12 nouns read aloud for 3 consecutive trials and each trial is followed by a recall test.
Time Frame: Open-label Baseline and Week 10
Population: FAS
Measure: Mean (Standard Deviation); unit: words recalled
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 73
words recalled | 0.7 (7.54)
Statistical Analysis 1: Comparison: SPD489 (Open-label Phase); Test type: Superiority or Other; p = 0.4312, t-test, 2 sided

20. Secondary Outcome: Change From Double-blind Randomization Baseline in HVLT-R Total Scores at Week 4 Double-blind Phase
Description: as for outcome 19
Time Frame: Double-blind Randomization Baseline and week 4 Double-blind Phase
Population: Randomized FAS
Measure: Least Squares Mean (Standard Error); unit: words recalled
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 31 | 31
words recalled | -1.5 (1.01) | 1.0 (1.01)
Statistical Analysis 1: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Test type: Superiority or Other; p = 0.0874, ANCOVA; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-5.4 to 0.4]

21. Secondary Outcome: Change From Open-label Baseline in University of California Performance-Based Skills Assessment, Brief Version (UPSA-B) Scores at Week 10 Open-label Phase, LOCF
Description: UPSA-B assesses skills in 5 areas of life functioning. It contains 2 subscales. Percentages correct on these 2 subscales are multiplied by 50. Thus, scores can range from 0 to 50 on each of these 2 subscales, and total scores can range from 0 to 100. Scores of 75 or higher are associated with independent living.
Time Frame: Open-label Baseline and week 10 Open-label Phase
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 83
Scores on a scale
  Total Skills | 6.2 (12.20)
  Communication Skills | 3.7 (8.56)
  Financial Skills | 2.5 (7.45)
Statistical Analysis 1: Comparison: SPD489 (Open-label Phase); Total Skills; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: SPD489 (Open-label Phase); Communication Skills; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided
Statistical Analysis 3: Comparison: SPD489 (Open-label Phase); Financial Skills; Test type: Superiority or Other; p = 0.0028, t-test, 2 sided

22. Secondary Outcome: Change From Double-blind Randomization Baseline in UPSA-B Scores at Week 4 Double-blind Phase
Description: as for outcome 21
Time Frame: Double-blind Randomization Baseline and Week 4 Double-blind Phase
Population: Randomized FAS
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 32 | 31
Scores on a scale
  Total Skills | -1.5 (1.35) | 0.0 (1.37)
  Communication Skills | -1.5 (1.14) | -0.6 (1.16)
  Financial Skills | -0.3 (0.83) | 0.9 (0.84)
Statistical Analysis 1: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Total Skills; Test type: Superiority or Other; p = 0.4637, ANCOVA; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-5.3 to 2.4]
Statistical Analysis 2: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Communication Skills; Test type: Superiority or Other; p = 0.6137, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-4.1 to 2.4]
Statistical Analysis 3: Comparison: SPD489 (Double-blind Phase) vs Placebo (Double-blind Phase); Financial Skills; Test type: Superiority or Other; p = 0.3482, ANCOVA; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-3.5 to 1.3]

23. Secondary Outcome: Change From Open-label Baseline in Behavioral Rating Inventory of Executive Function - Adult Version (BRIEF-A) T-scores at Week 10 Open-label Phase
Description: BRIEF-A is a validated 75-item questionnaire composed of three indexes (Global Executive Composite, Behavioral Recognition Index, and Metacognition Index). Items are rated 1 (never), 2 (sometimes), and 3 (often). Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Open-label Baseline and Week 10 Open-label Phase
Population: FAS
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 70
T-scores
  Global Executive Composite | -3.9 (13.29)
  Behavioral Recognition Index | -3.1 (12.89)
  Metacognition Index | -3.9 (13.12)
Statistical Analysis 1: Comparison: SPD489 (Open-label Phase); Global Executive Composite; Test type: Superiority or Other; p = 0.0174, t-test, 2 sided
Statistical Analysis 2: Comparison: SPD489 (Open-label Phase); Behavioral Recognition Index; Test type: Superiority or Other; p = 0.0461, t-test, 2 sided
Statistical Analysis 3: Comparison: SPD489 (Open-label Phase); Metacognition Index; Test type: Superiority or Other; p = 0.0146, t-test, 2 sided

24. Secondary Outcome: Change From Double-blind Randomization Baseline in BRIEF-A T-Scores at Week 4 Double-blind Phase
Description: as for outcome 23
Time Frame: Double-blind Randomization Baseline and Week 4 Double-blind Phase
Population: Randomized FAS
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 29 | 33
T-scores
  Global Executive Composite | -1.7 (1.19) | -1.2 (1.12)
  Behavioral Recognition Index | -0.9 (1.22) | -1.6 (1.14)
  Metacognition Index | -2.0 (1.26) | -0.7 (1.18)
Statistical Analysis 1: Comparison: SPD489 (Double-blind Phase); Global Executive Composite; Test type: Superiority or Other; p = 0.7418, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-3.8 to 2.7]
Statistical Analysis 2: Comparison: SPD489 (Double-blind Phase); Behavioral Recognition Index; Test type: Superiority or Other; p = 0.6429, ANCOVA; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-2.6 to 4.1]
Statistical Analysis 3: Comparison: SPD489 (Double-blind Phase); Metacognition Index; Test type: Superiority or Other; p = 0.4364, ANCOVA; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-4.8 to 2.1]

25. Secondary Outcome: Change From Open-label Baseline in Simpson Angus Scale (SAS) Total Score at Week 10 Open-label Phase
Description: SAS is a 10-item scale used to evaluate the presence and severity of extrapyramidal symptoms. The items are scored on a scale from 0 to 4 with item-specific definitions given for each point. Total scores range from 0 to 40. Lower scores indicate less impairment.
Time Frame: Open-label Baseline and Week 10 Open-label Phase
Population: SAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 70
Units on a scale | -0.01 (0.063)

26. Secondary Outcome: Change From Open-label Baseline in SAS Total Score at Week 4 of Double-blind Phase
Description: as for outcome 25
Time Frame: Open-label Baseline and Week 4 Double-blind Phase
Population: Randomized SAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 32 | 33
Units on a scale | 0.00 (0.093) | 0.00 (0.043)

27. Secondary Outcome: Change From Open-label Baseline in Barnes Akathisia Scale (BAS) Scores at Week 10 Open-label Phase
Description: BAS scale has objective, subjective, and global impression components of akathisia (motor restlessness that manifests itself with an inability to sit still or remain motionless). Objective and subjective components are rated on a scale from 0 (normal/absence) to 3 (severe) and are summed yielding a total score of 0 to 9. Global impression is rated on a scale from 0 (absent) to 5 (severe) with a total score ranging from 0 to 5. Lower scores indicate reduced restlessness.
Time Frame: Open-label Baseline and week 10 Open-label Phase
Population: SAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 70
Units on a scale
  Objective | 0.0 (0.17)
  Subjective | 0.0 (0.56)
  Global | 0.0 (0.36)

28. Secondary Outcome: Change From Open-label Baseline in BAS Scores at Week 4 of Double-blind Phase
Description: as for outcome 27
Time Frame: Open-label Baseline and Week 4 Double-blind Phase
Population: Randomized SAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 32 | 33
Units on a scale
  Objective | 0.0 (0.18) | -0.1 (0.24)
  Subjective | 0.0 (0.31) | -0.1 (0.65)
  Global | 0.0 (0.18) | -0.2 (0.44)

29. Secondary Outcome: Change From Open-label Baseline in Amphetamine Cessation Symptom Assessment (ACSA) Total Score at Week 10 Open-label Phase
Description: ACSA scale has 16 symptom items rated on a scale from 0 (not at all) to 4 (extremely) with a possible total score range of 0 to 64. Higher scores indicate greater withdrawal symptom severity.
Time Frame: Open-label Baseline and Week 10 Open-label Phase
Population: SAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 85
Units on a scale | -1.8 (9.69)

30. Secondary Outcome: Change From Double-blind Randomization Baseline in ACSA Total Score at Week 4 Double-blind Phase
Description: as for outcome 29
Time Frame: Double-blind Randomization Baseline and Week 4 Double-blind Phase
Population: Randomized SAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 29 | 29
Units on a scale | 0.4 (7.65) | -2.9 (8.75)

31. Secondary Outcome: Change From Open-label Baseline in Pittsburgh Sleep Quality Index (PSQI) Total Global Score at Week 10 Open-label Phase
Description: PSQI evaluates 7 areas of quality and pattern of sleep. Each area is rated on a scale from 0 (better) to 3 (worse) with a total score ranging from 0 to 21. Reduction in total scores are associated with better sleep quality.
Time Frame: Open-label Baseline and Week 10 Open-label Phase
Population: SAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 69
Units on a scale | -0.7 (3.15)

32. Secondary Outcome: Change From Open-label Baseline in PSQI Total Global Score at Week 4 of Double-blind Phase
Description: as for outcome 31
Time Frame: Open-label Baseline and Week 4 Double-blind Phase
Population: Randomized SAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 32 | 32
Units on a scale | 0.3 (3.01) | -1.7 (3.00)

33. Secondary Outcome: Change From Open-label Baseline in Calgary Depression Scale for Schizophrenia (CDSS) at Week 10 Open-label Phase
Description: CDSS is a 9-item scale to evaluate depression in subjects who have schizophrenia rated from 0 (absence of symptoms) to 3 (severe symptoms) with a total score range of 0 to 27. Lower scores indicate less depression.
Time Frame: Open-label Baseline and Week 10 Open-label Phase
Population: Safety Analysis Set (SAS) defined as all subjects who took at least 1 dose of open-label investigational product and for whom at least 1 follow-up safety assessment was made.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489 (Open-label Phase)
Number analyzed (Participants) | 70
Units on a scale | -0.7 (2.11)

34. Secondary Outcome: Change From Open-label Baseline in CDSS at Week 4 of Double-blind Phase
Description: as for outcome 33
Time Frame: Open-label Baseline and Week 4 of Double-blind Phase
Population: Randomized SAS defined as all subjects who took at least 1 dose of randomized investigational product and for whom at least 1 follow-up safety assessment was made.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 32 | 33
Units on a scale | -0.1 (2.34) | -0.7 (2.30)

ADVERSE EVENTS:
Description: Safety Analysis Set for both the Open-label and Double-blind Randomization Phases.
Groups:
- SPD489 (Open-label Phase); SPD489 (Double-blind Phase): Subjects receive either 20, 30, 40, 50, 60 or 70 mg of SPD489 (Lisdexamfetamine dimesylate) once-daily
- Placebo (Double-blind Phase): Subjects receive placebo once-daily
Arm/Group | SPD489 (Open-label Phase) | SPD489 (Double-blind Phase) | Placebo (Double-blind Phase)
Serious Adverse Events (participants affected / at risk) | 3/92 | 1/34 | 2/35
Other Adverse Events (participants affected / at risk) | 56/92 | 11/34 | 7/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPD489 (Open-label Phase) (N=92) | SPD489 (Double-blind Phase) (N=34) | Placebo (Double-blind Phase) (N=35)
Schizophrenia (Psychiatric disorders) | 1 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD489 (Open-label Phase) (N=92) | SPD489 (Double-blind Phase) (N=34) | Placebo (Double-blind Phase) (N=35)
Diarrhea (Gastrointestinal disorders) | 5 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 6 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 10 | 0 | 0
Dizziness (Nervous system disorders) | 8 | 0 | 0
Headache (Nervous system disorders) | 13 | 2 | 2
Insomnia (Psychiatric disorders) | 10 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 1
Fatigue (General disorders) | 4 | 2 | 1
Abdominal distention (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0 | 0
Nasopharyngitis (General disorders) | 2 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 0
Weight increased (Investigations) | 3 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Sedation (Nervous system disorders) | 2 | 0 | 0
Somnolence (Nervous system disorders) | 3 | 0 | 1
Agitation (Psychiatric disorders) | 3 | 1 | 0
Anxiety (Psychiatric disorders) | 4 | 1 | 0
Depressed mood (Psychiatric disorders) | 4 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Hernia (General disorders) | 0 | 0 | 1
Irritability (General disorders) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood pressure diastolic increased (Investigations) | 0 | 1 | 0
Blood prolactin increased (Investigations) | 0 | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.